CLINICAL TRIAL: NCT04618705
Title: The Role of the Gut Microbiome in Post-smoking Weight Gain
Brief Title: Gut Microbiome and Weight Gain After Smoking Cessation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: priority reasons
Sponsor: Eran Elinav (Other)
Responsible Party: Sponsor-Investigator, Eran Elinav, Principal Investigator, Host-Microbiome Interaction Research Group, Weizmann Institute of Science
Organization: Weizmann Institute of Science (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1093-1
Record Dates: First submitted 2020-10-21; First posted 2020-11-06 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-02

CONDITIONS: Smoking Cessation; Weight Gain
Keywords: Smoking cessation; Microbiome; Weight gain
MeSH Terms: conditions — Smoking Cessation; Weight Gain

STUDY DESIGN:
Intervention Model Description: Parallel non-randomized study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Participants who have not smoked for at least 10 years
- smoking group (No Intervention): Participants who have smoked cigarettes (at least 5 cigarettes per day) for at least 2 years.
- smoking cessation group (Experimental): Participants who have smoked cigarettes (at least 5 cigarettes per day) for at least 2 years and who are planning to quit smoking.
  Interventions: Behavioral: Smoking Cessation

INTERVENTIONS:
Behavioral: Smoking Cessation — Participants will start a smoking cessation program.
  Arms: smoking cessation group

SUMMARY:
Investigating the effect of smoking and smoking cessation on the intestinal microbial composition and function. The investigators wish to determine whether the alteration in gut microbiome drives the significant weight gain seen in humans after smoking cessation, and find the mechanism by which the gut microbiome contributes to this phenomenon.

DETAILED DESCRIPTION:
Cigarette smoking causes a variety of health problems, including cardiovascular disorders, cancer, pulmonary diseases, autoimmune diseases, premature birth, and certain birth defects. Health benefits of smoking cessation start very fast after the last smoke. However, smoking cessation has significant side effects including weight gain. Several theories have been proposed to explain weight gain after smoking cessation.

Microbiome research is an upcoming, extensively followed research field that has found unsuspected connections between human health and gut occupants. Many recent studies established important roles for the gut microbiome in regulating obesity, and metabolic diseases.

The general aim of this study is to investigate the effect of smoking and smoking cessation on the intestinal microbial composition and function.

This study follows 200 healthy participants who will be recruited according to their affiliation to one of three groups:

Group 1: Non-smokers for at least 10 years Group 2: Cigarette smokers that do not plan to quit. Group 3: Cigarette smokers who plan to quit smoking. Participants who are planning to quit cigarette smoking will be offered to join a program for smoking cessation. The study will start 8 days before cessation group volunteers will stop smoking and will continue for one year after. Participants of all groups will be followed-up for one year.

During the study, the participants will collect stool and oral samples which will be used for microbiota profiling. At every meeting anthropometric measurements, blood samples will be taken, and body composition performed. Participants will be connected to a continuous glucose monitor and will be asked to log a food diary using a designated mobile phone application.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smokers for at least 10 years, hereinafter 'control group'.
2. Cigarette smokers for at least 2 years, 5 or more cigarettes per day, that do not plan to quit hereinafter 'smoking group'.
3. Cigarette smokers for at least 2 years, 5 or more cigarettes per day, who plan to quit smoking hereinafter 'cessation group'.
4. Age - 18-70
5. BMI<28
6. Capable of working with the smartphone application in Hebrew or English.

Exclusion Criteria:

1. Consumption of antibiotics/oral antifungals/ probiotics 3 months before the first day of the experiment.
2. Constant consumption of drugs (cannabis etc..) in the last 2 years
3. Pregnancy in the last 6 months, breastfeeding, and active fertility treatments within the past year
4. Diagnosis of type 1 or type 2 diabetes
5. Chronic disease (infectious, autoimmune, endocrine, metabolic, neurodegenerative)
6. Cancer and recent anticancer treatment within the last 5 years
7. Neuro-psychiatric disorders
8. Coagulation disorders
9. Inflammatory bowel diseases (IBD)
10. Bariatric surgery within the last 5 years
11. BMI>28
12. Alcohol or substance abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Microbiome composition | 1 year
  Stool and oral samples

SECONDARY OUTCOMES:
Weight changes from baseline | 1 year
  Weight (Kg)
Blood glucose responses | 1 year
  Continuous glucose monitoring (CGM),

CONTACTS AND LOCATIONS:
Overall Officials: Eran Elinav, Prof, Principal Investigator — Weizmann Institute of Science

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and Health. The Health Consequences of Smoking-50 Years of Progress: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK179276/ PMID 24455788
- [Result] Benowitz NL. Cigarette smoking and cardiovascular disease: pathophysiology and implications for treatment. Prog Cardiovasc Dis. 2003 Jul-Aug;46(1):91-111. doi: 10.1016/s0033-0620(03)00087-2. No abstract available. PMID 12920702
- [Result] Grando SA. Connections of nicotine to cancer. Nat Rev Cancer. 2014 Jun;14(6):419-29. doi: 10.1038/nrc3725. Epub 2014 May 15. PMID 24827506
- [Result] Grumelli S, Corry DB, Song LZ, Song L, Green L, Huh J, Hacken J, Espada R, Bag R, Lewis DE, Kheradmand F. An immune basis for lung parenchymal destruction in chronic obstructive pulmonary disease and emphysema. PLoS Med. 2004 Oct;1(1):e8. doi: 10.1371/journal.pmed.0010008. Epub 2004 Oct 19. PMID 15526056
- [Result] Costenbader KH, Karlson EW. Cigarette smoking and autoimmune disease: what can we learn from epidemiology? Lupus. 2006;15(11):737-45. doi: 10.1177/0961203306069344. PMID 17153844
- [Result] Dahlin S, Gunnerbeck A, Wikstrom AK, Cnattingius S, Edstedt Bonamy AK. Maternal tobacco use and extremely premature birth - a population-based cohort study. BJOG. 2016 Nov;123(12):1938-1946. doi: 10.1111/1471-0528.14213. Epub 2016 Jul 14. PMID 27411948
- [Result] Hackshaw A, Rodeck C, Boniface S. Maternal smoking in pregnancy and birth defects: a systematic review based on 173 687 malformed cases and 11.7 million controls. Hum Reprod Update. 2011 Sep-Oct;17(5):589-604. doi: 10.1093/humupd/dmr022. Epub 2011 Jul 11. PMID 21747128
- [Result] Harris KK, Zopey M, Friedman TC. Metabolic effects of smoking cessation. Nat Rev Endocrinol. 2016 Nov;12(11):684. doi: 10.1038/nrendo.2016.171. Epub 2016 Sep 30. No abstract available. PMID 27688045
- [Result] Martinez de Morentin PB, Whittle AJ, Ferno J, Nogueiras R, Dieguez C, Vidal-Puig A, Lopez M. Nicotine induces negative energy balance through hypothalamic AMP-activated protein kinase. Diabetes. 2012 Apr;61(4):807-17. doi: 10.2337/db11-1079. Epub 2012 Feb 7. PMID 22315316
- [Result] Chen H, Hansen MJ, Jones JE, Vlahos R, Anderson GP, Morris MJ. Long-term cigarette smoke exposure increases uncoupling protein expression but reduces energy intake. Brain Res. 2008 Sep 4;1228:81-8. doi: 10.1016/j.brainres.2008.06.067. Epub 2008 Jun 26. PMID 18619427
- [Result] Ussar S, Griffin NW, Bezy O, Fujisaka S, Vienberg S, Softic S, Deng L, Bry L, Gordon JI, Kahn CR. Interactions between Gut Microbiota, Host Genetics and Diet Modulate the Predisposition to Obesity and Metabolic Syndrome. Cell Metab. 2015 Sep 1;22(3):516-530. doi: 10.1016/j.cmet.2015.07.007. Epub 2015 Aug 20. PMID 26299453
- [Result] Turnbaugh PJ, Ley RE, Mahowald MA, Magrini V, Mardis ER, Gordon JI. An obesity-associated gut microbiome with increased capacity for energy harvest. Nature. 2006 Dec 21;444(7122):1027-31. doi: 10.1038/nature05414. PMID 17183312
- [Result] Hur KY, Lee MS. Gut Microbiota and Metabolic Disorders. Diabetes Metab J. 2015 Jun;39(3):198-203. doi: 10.4093/dmj.2015.39.3.198. PMID 26124989